CLINICAL TRIAL: NCT04024839
Title: Comparison of Active Isolated Stretch and Post Isometric Relaxation for Hamstring Flexibility in Young Health Adults.
Brief Title: Comparison of Active Isolated Stretch and Post Isometric Relaxation for Hamstring Flexibility.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Jawad Naweed
Record Dates: First submitted 2019-07-13; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Hamstring Tightness
Keywords: Active isolated stretch; Active knee extension; Post isometric relaxation; Sit and reach test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Isometric Relaxation (Active Comparator): Post Isometric Relaxation was applied three times a week for the duration of three weeks.
  Interventions: Other: Post Isometric Relaxation
- Active Isolated stretch (Experimental): Active Isolated stretch was was applied three times a week for the duration of three weeks.
  Interventions: Other: Active Isolated Stretch

INTERVENTIONS:
Other: Active Isolated Stretch — In supine position, participant was asked to lock the knee and slowly lift leg using the quadriceps muscles. gentle assistance was given by the rope at the end of the movement, as the quadriceps muscles continue to move the leg. strech was applied for 2 sec and then release to starting position. two sets of 10 repetitions were performed.
  Arms: Active Isolated stretch
Other: Post Isometric Relaxation — In supine line, participant was asked to do SLR until resistance was met in hamstring muscles and then was asked to do isometric contraction (10-20% of maximum) for 5 - 10 sec and inhale. After this, patient was asked to exhale while doing so gentle stretch was applied till the new barrier. Starting from this new barrier, the procedure was repeated 2 - 3 times.
  Arms: Post Isometric Relaxation

SUMMARY:
This study was intended to compare the immediate, short term and long term effects of active isolated stretch versus post isometric relaxation on hamstring flexibility in young healthy adults.35 students were assigned randomly into two groups with 17 and 18 in each group. Group A was given post isometric relaxation while Group B was Active isolated stretch. 22.2 year male and female students with tight hamstring were included while any neurological and orthopedic disorder were excluded. Active Isolated Stretch and Post Isometric Relaxation at baseline, after first and final exercise session were calculated immediate and short term effects while long term effects were calculated after two weeks of final session.

DETAILED DESCRIPTION:
Hamstring muscle is present on posterior region of thigh starting from gluteal region and ending in popliteal fossa. Hamstring has three muscles biceps femoris, semitendinosus and semimembranosus causing flexion at knee joint and help in extension of thigh. Biceps femoris further consists of two heads (long and short head). Long head is supplied by tibial part of the sciatic nerve, while short head is supplied by the common peroneal part of the sciatic nerve. Muscles such as gastro-soleus, tibialis posterior, rectus femoris, iliopsoas, tensor fasica lata, the hamstrings and hip adductors are more likely to be tightened in lower limbs. Muscle tightness can cause the muscle shortness and does not allow full passive or active range of motion. Full active and passive range of motion is only achieved when muscle is flexible.

Tightness of hamstring muscle can occur due to many reasons like injury to the muscle, prolonged sitting hours which are part of different jobs and educational setups. This tightness could lead to strain of the hamstrings, which is the most common occurring injury of the lower limbs. Moreover, hamstring tightness is also correlated with low back pain and lumbar dysfunction. Massage and stretching relax the tightened muscles but cannot normalize the tone or improve their coordination. To achieve this, investigator retrained muscle memory by actively using those respective muscles. Simple stretching of different muscle groups especially hamstrings has been found to improve the extensibility and length of shortened muscles.

Additionally, muscle Energy Techniques (MET) and their related post-isometric relaxation techniques have demonstrated better results in improving flexibility of the tightened muscles. Muscle Energy Techniques are used in soft tissue pathologies in which the patient performs active muscle contraction in specific positions and in specific direction against a force applied by the therapist. The therapist guides and controls the movement with instruction. These are manual techniques that use contraction of the specific muscles and are found to be effective in increasing flexibility of the muscles and improving range of motion. The underlying mechanism through which improvement in extensibility and length occurs is yet unclear and thought to be attributed to both mechanical as well as neurological factors. Firstly MET techniques applied to increase extensibility of the muscles typically involves following steps: stretching the muscle to the limit of barrier or person's tolerance, secondly the person performs an active isometric contraction of the muscle being stretched against a controlled resistance provided by the therapist, additionally the person relaxes the muscle being stretched while the therapist continues holding the stretched position, furthermore the therapist takes up the new range produced by muscle and lengthens it up to a new barrier, and this whole procedure is repeated again according to defined guidelines. The MET techniques can be modified with variations in different components such as force of contraction, duration of the contraction, duration of the stretch and repetitions. This whole process results in increased range of motion and improves flexibility.

Post Isometric Relaxation (PIR) is a type of MET that relaxes the tight muscles with avoidance of initiating stretch reflex. This in turn results in reduced spasm and improved ROM. The relaxation is induced due to isometric contraction of the muscles with facilitation and inhibition. Active Isolated Stretch (AIS) is another type of stretching in which specific movement is performed for a specific muscle with assistance from a therapist or self-assisted (with rope or a band) and those particular movements are repeated again and again to induce a relaxation phenomenon in muscles, fascia and connective tissues. In AIS, movements are monitored carefully to avoid producing any stretch reflex .

A single blind randomized control study was done in Islamabad federal college Islamabad with the duration of 6 months from Jan 2018 to July 2018.the calculated sample size was 35 students (17 in group A and 18 in group B) through open epi . Non probability random sample selection method was used on the behalf of inclusion and exclusion criteria. 22.2+ 2.02 year male and female students of DPT with tight hamstring were included while hamstring injury and any neurological or orthopedic disorder were excluded. The study was approved by the Ethical and Research Committee, and all participants signed the informed consents. Group A was given post isometric relaxation while Group B was given Active isolated stretch for a period of 3 weeks. Outcome measures were assessed at baseline, after first and final exercise session to estimate immediate and short term effects while long term effects were calculated after two weeks of final session of interventions. Semi structured questionnaire was used for subjective and objective assessment. AKE score, sit and reach test score and Lower Extremity Functional Scale questionnaire was used to assess lower extremity functional activities. Sit and reach test was also used to measure hamstring length.

ELIGIBILITY:
Inclusion Criteria:

- Tight hamstring (Inability to achieve greater than 160° of knee extension with hip at 90° of flexion).

Exclusion Criteria:

* Having hamstring injury in past 6 months
* Having any neurological or orthopedic disorder effecting low back and lower limbs.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Active knee extension score | Upto 5 weeks
  The Active Knee Extension Test is used to assess hamstring muscle length and the range of active knee extension in the position of hip flexion. The measurement unit is degrees on the goniometer.

SECONDARY OUTCOMES:
Sit and reach test | Upto 5 weeks
  The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles. The score is recorded to the nearest centimeter or half inch as the distance reached by the hand.

OTHER OUTCOMES:
Lower extremity functional scale | after 2 weeks of intervention
  The objective of the Lower Extremity Functional Scale (LEFS) is to measure "patients' initial function, ongoing progress, and outcome" for a wide range of lower-extremity conditions. Patients select an answer from the following scale for each activity listed:
  Extreme Difficulty or Unable to Perform Activity, Quite a Bit of Difficulty, Moderate Difficulty, A Little Bit of Difficulty, No Difficulty,
  The patient's score is tallied at the bottom of the page. The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feland JB, Myrer JW, Schulthies SS, Fellingham GW, Measom GW. The effect of duration of stretching of the hamstring muscle group for increasing range of motion in people aged 65 years or older. Phys Ther. 2001 May;81(5):1110-7. PMID 11319936
- [Background] Handel M, Horstmann T, Dickhuth HH, Gulch RW. Effects of contract-relax stretching training on muscle performance in athletes. Eur J Appl Physiol Occup Physiol. 1997;76(5):400-8. doi: 10.1007/s004210050268. PMID 9367279
- [Background] Smith M, Fryer G. A comparison of two muscle energy techniques for increasing flexibility of the hamstring muscle group. J Bodyw Mov Ther. 2008 Oct;12(4):312-7. doi: 10.1016/j.jbmt.2008.06.011. Epub 2008 Aug 6. PMID 19083689
- [Background] van Gent RN, Siem D, van Middelkoop M, van Os AG, Bierma-Zeinstra SM, Koes BW. Incidence and determinants of lower extremity running injuries in long distance runners: a systematic review. Br J Sports Med. 2007 Aug;41(8):469-80; discussion 480. doi: 10.1136/bjsm.2006.033548. Epub 2007 May 1. PMID 17473005